CLINICAL TRIAL: NCT00348634
Title: The Effects of Tegaserod on Orocecal Transit in Elderly Patients With Chronic Constipation
Brief Title: Effect of Tegaserod on Orocecal Transit in Elderly Chronic Constipation Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated early due to regulatory action suspending tegaserod use in 2007
Sponsor: Novartis (Industry)
Collaborators: Temple University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919EUS51
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Constipation
Keywords: Constipation, Tegaserod, orocecal transit, colonic transit, gastric emptying
MeSH Terms: conditions — Constipation | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study will evaluate the effects of tegaserod on orocecal and colonic transit in patients over 65 years with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Male & Females aged 65 and older
* Patients must meet the criteria for chronic idiopathic constipation for at least 12 weeks
* Patients must have had a colonoscopy within the past 5 years
* Patients must pass a balloon expulsion test at screening
* Patients must be able to comply and understand the use of a diary

Exclusion Criteria:

* Patients with a clinically significant medical condition that would interfere with the patient completing the trial
* Patients with loose stools at least once per week
* Patients with IBS
* Known allergies to the same class of drug and/or allergies to eggs
* Patients who require the use of manual maneuvers to have a bowel movement

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Orocecal transit: Time of radioactive marker to reach the cecum using scintigraphy

SECONDARY OUTCOMES:
Whole gut transit and stomach emptying: Following 2 weeks of treatment, the rate of transit of food through the colon and stomach will be measured using scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Henry Parkman, MD, Study Chair — Temple; William Chey, MD, Study Chair — University of Michigan
Locations (3):
- United States (3):
  - Arkansas Gastroenterology, PA, North Little Rock, Arizona
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Temple University Hospital, Philadelphia, Pennsylvania